CLINICAL TRIAL: NCT02316665
Title: Effect of Continuous Positive Airway Pressure Treatment on Nocturnal Glycemia of Patients Having Type 1 Diabetes and Sleep Apnea Syndrome: a Randomized Controlled Trial
Brief Title: Effect of Sleep Apnea Treatment on Type 1 Diabetes
Acronym: DIADEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Société francophone de pneumologie de langue francaise (Unknown); ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-A006336-40
Record Dates: First submitted 2014-09-22; First posted 2014-12-15 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes; Sleep Apnea Syndrome
Keywords: Type 1 diabetes; Sleep apnea syndrome; Nocturnal glycemia; Continuous glucose monitoring system; Continuous positive airway pressure; Sleep habits
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous positive airway pressure (Experimental): Patients will receive continuous positive airway pressure during three months
  Interventions: Device: continuous positive airway pressure
- Sham-continuous positive airway pressure (Sham Comparator): Patients will receive sham-continuous positive airway pressure during 3 months
  Interventions: Device: Sham-continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — continuous positive airway pressure treatment during three months with adherence recording
  Arms: continuous positive airway pressure
Device: Sham-continuous positive airway pressure — Sham-continuous positive airway pressure during three months with adherence recording
  Arms: Sham-continuous positive airway pressure

SUMMARY:
Hypothesis: To address the role of continuous positive airway pressure (CPAP)on nocturnal glycemia in patients having type 1 diabetes and sleep apnea syndrome.

Investigators make the hypothesis that sleep apnea syndrome impacts nocturnal glycemia in type 1 diabetic patients and that continuous positive airway pressure treatment will permit to improve the nocturnal glycemic profile.

Study design: Adult patients with type 1 diabetes will be recruited for an extensive study of sleep habits and assessment of sleep breathing disorders. When patients will present with severe sleep apnea syndrome (apnea-hypopnea index above 30 events/hour) and insufficient glycemic control (HbA1c > 7.5%), they will be randomized in continuous positive airway pressure treatment or sham-continuous positive airway pressure treatment group for three months.

Main outcome: Nocturnal glycemic control will be assessed for 5 days before and after three months of the allocated treatment.

DETAILED DESCRIPTION:
Quality of clinical study procedures will be checked by on-site audit.

Patient self-reported past medical history will be checked by reviewing medical records.

Paper case report forms will be used.

For the baseline extensive study of sleep habits, the following data are recorded:

* Self-reported sleep diary (7 days)
* Actimetric device (7 days)
* Munich Chronotype Questionnaire
* 24h-dietary recall
* Salivary collections every 30 minutes between 7:30 pm and 22:00 pm on one night to address the dim light melatonin onset.
* Other questionnaires: Job strain questionnaire, EPICES (precarity questionnaire) and DQOL (diabetes related quality of life)
* Nocturnal oxymetry

Blood measurements: HbA1c, lipidic profile, microalbuminuria, creatinin

After baseline assessment, patients having an abnormal nocturnal oximetry will be explored by polysomnography in order to detect a sleep apnea syndrome.

Investigators anticipate, based on a previous pilot study of our group ("Borel" Diab Med 2010), that 30% of screened patients will present with sleep apnea.

If patients present with severe sleep apnea (IAH > 30 events/hour) and HbA1c > 7.5%, they will be randomized for the intervention.

Sample size: based on a previous study by "Pallayova" et al. in patients having type 2 diabetes, investigators anticipate a difference between groups of 1.3 (SD 2.07) for the mean nocturnal glycemia. For a alpha threshold of 5% and a study power of 80%, the study should include 32 patients in each group. Taking in account a possible 25% of dropout the study will need to include 40 patients by randomized arm to demonstrate an effect.

Statistical analysis: An intention-to-treat analysis will be performed. Missing data for the continuous positive airway pressure group will be replaced by the median value at three-month of the sham-continuous positive airway pressure group and reciprocally.

In a second analysis, a per-protocol analysis will be performed limited to patients having completed their treatment in allocated group and having an adherence to continuous positive airway pressure or sham-continuous positive airway pressure treatment for more than 4-hours a night.

Normality of data will be checked by Kurtosis and Skewness tests. The significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with type 1 diabetes

Exclusion Criteria:

* Pregnant women
* Patient with acute metabolic disorders during the past three months
* Shift workers
* Institutionalized patient
* Enteral and parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change in mean nocturnal glycemia | 3 months
  Measured from continuous glycemic monitoring system

SECONDARY OUTCOMES:
Change in blood pressure | 3 months
  24h ambulatory blood pressure monitoring
Change in the variability of nocturnal glycemia | 3months
  Measured on nighttime recording of continuous glycemic monitoring system
Change in HbA1c | 3 months
Changes in sleep duration after intervention | 3 months
  Actimetry
Change in mean systolic blood pressure after intervention | 3 months
  Self-monitoring blood pressure and heart rate device, at home
Chang in sleep timing after intervention | 3 months
  Actimetry
Change in daily activity after intervention | 3 months
  Actimetry
Change in mean diastolic blood pressure after intervention | 3 months
  Self-monitoring blood pressure and heart rate device, at home
Change in mean heart rate after intervention | 3 months
  Self-monitoring blood pressure and heart rate device, at home

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD PhD, Principal Investigator — HP2 INSERM U1042 laboratory, France
Locations (1):
- Grenoble University hospital, Grenoble, France